CLINICAL TRIAL: NCT02491489
Title: A Comparison of the Effects of Glenohumeral Mobilization on Rotator Cuff Activity in Normal and Painful Shoulders
Brief Title: Activity of the Rotator Cuff During Glenohumeral Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCEMG
Record Dates: First submitted 2015-06-29; First posted 2015-07-08 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2015-06

CONDITIONS: Shoulder Pain
Keywords: Manual therapy
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Painful shoulders (Experimental): Subjects with shoulder pain undergoing glenohumeral mobilization
  Interventions: Other: Glenohumeral mobilization
- Normal shoulders (Active Comparator): Subjects without shoulder pain undergoing glenohumeral mobilization
  Interventions: Other: Glenohumeral mobilization

INTERVENTIONS:
Other: Glenohumeral mobilization — Participants will then be placed supine on a standard plinth. The investigators will then proceed to provide a mobilizing force to the participant's glenohumeral joints. Each of two investigators will, in sequence perform a 15 second longitudinal distraction, followed by a 15 second posteriorly directed glenohumeral glide with the shoulder placed in the open pack resting position (~50 degrees abduction, slight horizontal adduction, external rotation).

SUMMARY:
Shoulder pain is one of the most common musculoskeletal conditions treated by physical therapists. One common treatment is passive glenohumeral joint accessory mobilization, which is the application of a therapist generated force to move the humeral head (ball) on the glenoid (socket) of the shoulder to improve motion and decrease pain. It is generally accepted that these mobilizations do not elicit active muscular contractions of the surrounding musculature. However, there is very little literature to support this assumption, and a preliminary PubMed search utilizing the terms "shoulder"," mobilization", and "EMG" returned zero relevant references. Therefore, the investigators plan to utilize surface electromyography (EMG), a non-invasive assessment tool, to objectively measure the activity of the rotator cuff muscles (the muscles that surround the shoulder and provide stability to the joint) during various grades(levels of force and amplitude of movement) of glenohumeral mobilization ( a standard of care treatment). It is also unknown if subjects pain levels impact the level of rotator cuff activity. To investigate these questions, the investigators will collect EMG data while performing mobilizations on a total of 20 subjects, divided into two groups: 10 pain free shoulders and 10 painful shoulders. Data analysis will then include descriptive analysis, estimates of effect size, and analysis for between group differences.

The investigators hypothesize that there will be significant differences in muscular activity between groups related to the presence of shoulder pain.

DETAILED DESCRIPTION:
Following informed consent, all participants will be assessed in a private EMG lab setting. After exposing the posterior shoulder girdle, the areas of the upper trapezius, supraspinatus, and infraspinatus will be cleaned using a cloth alcohol prep pad, and the skin at the area of electrode placement will be vigorously abraded for 5 seconds. A previously calibrated (per Delsys system protocol) Delsys mini-wireless electrode will then be placed at the appropriate location over each muscle as described by Criswell. These electrodes will be securely taped in place using specialized tape as specified by the manufacturer.

Once electrode placement is complete, each participant will first undergo a standardizing reference contraction of each muscle group. For the upper trapezius, this will consist of 1) a 9 second shrug,2) 9 second elevation of the arm to 90 degrees in the empty can position, and 3) a side lying external rotation of the shoulder to 90 degrees. The middle 3 seconds of each trial will be used to record the average electrical activity of each muscle during voluntary contraction.

Participants will then be placed supine on a standard plinth. The investigators will then proceed to provide a mobilizing force to the subject's glenohumeral joints. Each of two investigators will, in sequence perform a 15 second longitudinal distraction, followed by a 15 second posteriorly directed glenohumeral glide with the shoulder placed in the open pack resting position (~50 degrees abduction, slight horizontal adduction, external rotation). The middle 5 seconds will be captured for mean electrical activity at each of the three previously identified muscles. Following completion of the mobilizations by the second investigator, the electrodes will be removed, and the subject's participation will be complete.

Data analysis will include basic subject demographics such as age, gender, and handedness. Tests of between group difference will be analyzed for each mobilization and tester condition. Data will be analyzed comparing mean EMG values during mobilization compared to the active contraction using the reference voluntary contraction (RVC) method, as this has been shown be a more accurate comparator for low levels of muscle activity.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals and subjects with shoulder pain
* ages 18-64
* all subjects must be ambulatory, able to transfer onto a standard treatment plinth, and able to tolerate lying supine (on their back) for a minimum of 15 minutes.

Exclusion Criteria:

* recent (6 months) shoulder surgery
* shoulder replacement on the involved side
* any history of shoulder fractures
* active cancer or metastatic disease
* coagulation disorders
* current pregnancy
* rheumatoid arthritis
* active litigation for current injury
* active workman's compensation for current injury
* osteoporosis

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
EMG activity of the rotator cuff using % reference voluntary contraction method | EMG data will be collected simultaneously during the intervention
  EMG activity collected during the intervention will be compared to the baseline reference contractions.